CLINICAL TRIAL: NCT07346534
Title: Reinforced Versus Conventional Anastomosis in Laparoscopic Low Rectal Cancer Resection: A Comparative Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Feng-Min, Investigator assistant, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25K50
Record Dates: First submitted 2025-07-16; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Low Rectal Cancer; Rectal Neoplasms; Colorectal Cancer
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reinforced Anastomosis with 8-10 Interrupted Sutures (Experimental): Patients in this group will undergo laparoscopic low anterior resection (Dixon procedure) for low rectal cancer, followed by reinforcement of the anastomosis using 8-10 interrupted seromuscular sutures circumferentially around the stapled anastomotic site. The reinforcement is intended to enhance anastomotic integrity and reduce the risk of leakage.
  Interventions: Procedure: Reinforced Anastomotic Suturing (8-10 Interrupted Sutures)
- Conventional Dixon Procedure (Active Comparator): Patients in this group will undergo standard laparoscopic low anterior resection (Dixon procedure) for low rectal cancer without additional reinforcement of the anastomosis. The anastomosis will be performed using a circular stapler alone, as per conventional practice.
  Interventions: Procedure: Conventional Laparoscopic Dixon Procedure

INTERVENTIONS:
Procedure: Reinforced Anastomotic Suturing (8-10 Interrupted Sutures) — After completing the laparoscopic low anterior resection (Dixon procedure) for low rectal cancer, the surgeon performs additional reinforcement of the colorectal anastomosis. This is done by placing 8 to 10 interrupted seromuscular sutures circumferentially around the anastomotic site. The goal of this reinforcement is to enhance anastomotic stability, promote healing, and reduce the risk of anastomotic leakage.
  Arms: Reinforced Anastomosis with 8-10 Interrupted Sutures
Procedure: Conventional Laparoscopic Dixon Procedure — Patients undergo standard laparoscopic low anterior resection (Dixon procedure) for low rectal cancer. The colorectal anastomosis is performed using a circular stapler without any additional suturing or reinforcement. This represents the conventional surgical approach widely used in clinical practice.
  Arms: Conventional Dixon Procedure

SUMMARY:
Study Description This prospective, controlled clinical study aims to compare the clinical outcomes of reinforced anastomosis using 8-10 interrupted sutures versus the conventional Dixon procedure in patients undergoing laparoscopic low anterior resection for low rectal cancer. Anastomotic leakage remains one of the most significant postoperative complications following low rectal cancer surgery, particularly in laparoscopic procedures due to limited tactile feedback and maneuverability in the pelvic cavity.

Reinforcement of the anastomotic site through additional interrupted suturing may provide better mechanical strength and improved healing, potentially reducing the incidence of anastomotic leakage and related morbidities. In this study, eligible patients will be assigned to receive either a conventional laparoscopic Dixon procedure or the same procedure with added reinforcement of the anastomosis using 8-10 interrupted sutures circumferentially.

Perioperative outcomes including the rate of anastomotic leakage, postoperative complications, operation time, length of hospital stay, return of bowel function, and quality of life will be assessed and compared between the two groups. The study seeks to provide evidence for optimizing surgical techniques in low rectal cancer treatment and improving patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years.
2. Diagnosed with low rectal adenocarcinoma located within 7 cm from the anal verge by colonoscopy and biopsy.
3. Scheduled for elective laparoscopic low anterior resection (Dixon procedure).
4. Clinical stage I-III (based on preoperative imaging, e.g., MRI/CT) without distant metastasis.
5. Adequate organ function (hematologic, hepatic, renal) to tolerate surgery.
6. Provided written informed consent and willing to comply with study procedures and follow-up.

Exclusion Criteria:

1. Presence of synchronous distant metastases or other malignancies.
2. History of prior pelvic radiotherapy or major pelvic surgery.
3. Severe uncontrolled comorbidities (e.g., severe cardiovascular, respiratory, hepatic or renal insufficiency).
4. Emergency surgery indication (e.g., bowel obstruction, perforation).
5. Pregnancy or breastfeeding.
6. Known allergy or contraindication to anesthesia or surgical materials used.
7. Participation in another interventional clinical trial within the last 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Anastomotic Leakage | Within 30 days postoperatively
  Defined as clinically significant leakage confirmed by radiological or surgical evidence, classified according to International Study Group of Rectal Cancer (ISREC) criteria.

SECONDARY OUTCOMES:
Postoperative Complication Rate | Up to 30 days after surgery
  Incidence of Clavien-Dindo grade II or higher complications.
Operation Time | During the surgical procedure
  Total duration of surgery from skin incision to skin closure.
Length of Postoperative Hospital Stay | From date of surgery through date of discharge, up to 30 days
  Number of days from surgery to hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No